CLINICAL TRIAL: NCT06638567
Title: Postoperative Glucose Control with a Basal Bolus Versus Sliding Scale Insulin Regimen and Its Effect on the Incidence of Surgical Site Infections in People with Type 2 Diabetes Mellitus.
Brief Title: Postoperative Basal Bolus or Sliding Scale Insulin Regimen in DM2 and Its Effect on Surgical Site Infections.
Acronym: GUIDE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abraham Hulst, MD, PhD (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor-Investigator, Abraham Hulst, MD, PhD, Clinical investigator, anesthesiologist, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GUIDE trial
Record Dates: First submitted 2024-03-10; First posted 2024-10-15 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus, Type 2; Surgical Site Infection
Keywords: Diabetes Mellitus; Basal bolus regimen; Surgical site infections; Sliding scale; Insulin regimen
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Surgical Wound Infection; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Multicenter, matched, cluster-randomised
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Basal Bolus (Experimental): Patients daily dose of insulin is calculated by their treatment team: In insulin naive patients 0.4-0.5IU/kg and 0,3IU/kg for patients aged>70 or patients with impaired kidney function with an estimated glucose filtration rate <60ml/min and 80-100% of own insulin for insulin-users. They receive half of this daily dose in long-acting insulin once a day. The other half of their total daily dose of insulin is provided as short-acting mealtime insulin. This short-acting insulin is administered before each meal. When needed, extra insulin can be given when needed.
  The measurements of blood glucose values are before each meal and at bedtime (4x/day).
  Interventions: Other: Basal bolus insulin regimen
- Sliding Scale (No Intervention): Short-acting insulin is administered when blood glucose value is above 10,0 mmol/L according to a standardized dosage schedule. The measurements of blood glucose values are before each meal and at bedtime (4x/day).

INTERVENTIONS:
Other: Basal bolus insulin regimen — Combination of long-acting and short-acting insulin in a proactive schedule for achieving better blood glucose values postoperatively
  Arms: Basal Bolus

SUMMARY:
A multicentre, matched-pair, cluster randomised controlled superiority trial to investigate the effect of a proactive basal bolus insulin regimen compared to the reactive sliding scale insulin regimen, targeting a glucose level of 3.9-10.0 mmol/L, to reduce the number of surgical site infections within the first 30 days postoperatively in adult patients with diabetes mellitus type 2.

DETAILED DESCRIPTION:
People with type 2 diabetes mellitus (PWT2D) are at increased risk of postoperative complications, especially surgical site infections (SSI).

The aim of this study to reduce SSI in PWT2D by implementing a proactive basal-bolus insulin regimen, compared to the reactive sliding scale regimen.

Adult patients with type 2 diabetes will be included in this multi-centre study.

Participants will receive a blind CGM, i.e. glucose data are masked for the participants and study team, from admission to the ward until discharge from the hospital. In addition, all participants are asked to complete several questionnaires 30 days after surgery.

Both regimens are currently used in clinical practice. Therefore, there is no additional trial-related burden depending on the intervention group allocation.

Participants will be monitored intensively and insulin dosage will be adjusted adequately to the measured glucose values by the treatment team.

The sample size is based on the SSI incidence rates. Wards are matched into pairs with comparable baseline incidence rates and in each pair, one ward will be randomly assigned to the intervention group; the other serves as the control. 18 wards from 8 participating centres are planned to be recruited, this translates to 9x2x56=1008 evaluable participants.

Keywords:

Diabetes mellitus, basal bolus, sliding scale, insulin regimen, surgical site infections

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or older
* Diagnosed with type 2 diabetes mellitus
* Undergoing gastointestinal or vascular surgery
* Admitted to one of the participating surgical wards
* Expected duration of stay at least one overnight stay
* Willing and able to provide informed consent

Exclusion Criteria:

* Diagnosed with type 1 diabetes mellitus
* Female of child-bearing potential who is pregnant or breastfeeding.
* Undergoing complete pancreatectomy
* Undergoing bariatric surgery
* Patients using a continuous insulin pump at home
* Patients undergoing a necrotectomy/wound debridement from a pre-existent wound.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1008 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Surgical site infection | Until 30 days after surgery
  Incidence of postoperative surgical site infection, according to the criteria of the centres of disease control (CDC) for superficial incisional SSI, deep incisional SSI and organ / space SSI.
  SSIs will be measured at 30 days postoperatively via BLUEBELLE questionnaire, diagnosis by surgeon during standard postoperative visit at the surgery clinic 3-5 weeks after surgery and chart review.

SECONDARY OUTCOMES:
Postoperative hospital-acquired infections (non-SSI) | Recorded at 30 days postoperatively
  Incidence of hospital-acquired infections, other than surgical site infections
Length of stay in the hospital (LoS-Hos) | Recorded at 30 days postoperatively
  Length of stay in the hospital, measured in days from admission to discharge from the hospital.
Hospital readmission | Recorded 30 days postoperatively
  Rate of hospital readmissions within 30 days after surgery
Days at home (DAH30) | Recorded 30 days postoperatively
  Patient-reported number of days at home after surgery, between 0 and 30.
Postoperative disability | Recorded 30 days postoperatively
  Patient-reported level of disability 30 days after surgery, using the WHODAS-2.0 questionnaire. Summarized in a score between 0-100.
Quality of life (QoL) after surgery | Recorded 30 days postoperatively
  Patient-reported health-related quality of life 30 days after surgery, using the EuroQol 5D5L questionnaire, summarized in a score between 0 and 1.
Glucose 2 | Measured 4 times a day, until discharge from the hospital, up to 30 days.
  Incidence of grade 2 hypoglycemia, a blood glucose below 3.0mmol/L.
Glucose 3 | Measured 4 times a day, until discharge from the hospital, up to 30 days.
  Incidence of grade 1 hyperglycemia, a blood glucose above 10.0mmol/L.
Glucose 4 | Measured 4 times a day, until discharge from the hospital, up to 30 days.
  Incidence of grade 2 hyperglycemia, a blood glucose above 14.0mmol/L.
CGM1 | Measured with a 5-minute interval, until discharge from the hospital, up to 30 days.
  Percentage of time within glycaemic target range (3.9-10.0 mmol/L) per day and over hospital admission. This is measured with the continuous glucose monitor (CGM).
CGM2 | Measured with a 5-minute interval, until discharge from the hospital, up to 30 days.
  Percentage of time below glycaemic target range (<3.9mmol/L) per day and over hospital admission. This is measured with the continuous glucose monitor (CGM).
CGM3 | Measured with a 5-minute interval, until discharge from the hospital, up to 30 days.
  Percentage of time above glycaemic target range (>10.0mmol/L) per day and over hospital admission. This is measured with the continuous glucose monitor (CGM).
Cost-effectiveness 1 | Until 30 days after surgery
  The cost-effectiveness of the basal bolus insulin regimen compared to the sliding scale regimen, considering the costs per prevented of SSI in a cost-effectiveness analysis.
Cost-effectiveness 2 | Up to 30 days after surgery.
  The number of quality adjusted life years (QALYs) gained after a cost-utility analysis.
Protocol adherence | During the hospital stay, until discharge
  The adherence to the protocol until discharge from the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Sarah E. Siegelaar, MD, PhD, Principal Investigator — Amsterdam UMC, location AMC
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Complete data collection methods and results will be shared with other researchers upon a formal request made to the principal investigator including a detailed motivation for the request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: One year after reviewed publication of the primary results
Access Criteria: Official request to the principal investigator

REFERENCES:
- [Background] Kao LS, Phatak UR. Glycemic control and prevention of surgical site infection. Surg Infect (Larchmt). 2013 Oct;14(5):437-44. doi: 10.1089/sur.2013.008. Epub 2013 Oct 10. PMID 24111757
- [Background] Kotagal M, Symons RG, Hirsch IB, Umpierrez GE, Dellinger EP, Farrokhi ET, Flum DR; SCOAP-CERTAIN Collaborative. Perioperative hyperglycemia and risk of adverse events among patients with and without diabetes. Ann Surg. 2015 Jan;261(1):97-103. doi: 10.1097/SLA.0000000000000688. PMID 25133932
- [Background] Polderman JA, Van Velzen L, Wasmoeth LG, Eshuis JH, Houweling PL, Hollmann MW, Devries JH, Preckel B, Hermanides J. Hyperglycemia and ambulatory surgery. Minerva Anestesiol. 2015 Sep;81(9):951-9. Epub 2015 Jan 16. PMID 25592489
- [Background] de Vries FE, Gans SL, Solomkin JS, Allegranzi B, Egger M, Dellinger EP, Boermeester MA. Meta-analysis of lower perioperative blood glucose target levels for reduction of surgical-site infection. Br J Surg. 2017 Jan;104(2):e95-e105. doi: 10.1002/bjs.10424. Epub 2016 Nov 30. PMID 27901264
- [Background] Umpierrez GE, Smiley D, Jacobs S, Peng L, Temponi A, Mulligan P, Umpierrez D, Newton C, Olson D, Rizzo M. Randomized study of basal-bolus insulin therapy in the inpatient management of patients with type 2 diabetes undergoing general surgery (RABBIT 2 surgery). Diabetes Care. 2011 Feb;34(2):256-61. doi: 10.2337/dc10-1407. Epub 2011 Jan 12. PMID 21228246
- [Background] de Lissovoy G, Fraeman K, Hutchins V, Murphy D, Song D, Vaughn BB. Surgical site infection: incidence and impact on hospital utilization and treatment costs. Am J Infect Control. 2009 Jun;37(5):387-397. doi: 10.1016/j.ajic.2008.12.010. Epub 2009 Apr 23. PMID 19398246
- [Background] Phillips VL, Byrd AL, Adeel S, Peng L, Smiley DD, Umpierrez GE. A Comparison of Inpatient Cost Per Day in General Surgery Patients with Type 2 Diabetes Treated with Basal-Bolus versus Sliding Scale Insulin Regimens. Pharmacoecon Open. 2017;1(2):109-115. doi: 10.1007/s41669-017-0020-9. Epub 2017 Apr 21. PMID 28660256
- [Background] Koek MBG, van der Kooi TII, Stigter FCA, de Boer PT, de Gier B, Hopmans TEM, de Greeff SC; Burden of SSI Study Group. Burden of surgical site infections in the Netherlands: cost analyses and disability-adjusted life years. J Hosp Infect. 2019 Nov;103(3):293-302. doi: 10.1016/j.jhin.2019.07.010. Epub 2019 Jul 19. PMID 31330166
- [Background] Fowler AJ, Wahedally MAH, Abbott TEF, Smuk M, Prowle JR, Pearse RM, Cromwell DA. Death after surgery among patients with chronic disease: prospective study of routinely collected data in the English NHS. Br J Anaesth. 2022 Feb;128(2):333-342. doi: 10.1016/j.bja.2021.11.011. Epub 2021 Dec 20. PMID 34949439
- [Background] Dungan KM, Braithwaite SS, Preiser JC. Stress hyperglycaemia. Lancet. 2009 May 23;373(9677):1798-807. doi: 10.1016/S0140-6736(09)60553-5. PMID 19465235
- [Background] Lai J, Li Q, He Y, Zou S, Bai X, Rastogi S. Glycemic Control Regimens in the Prevention of Surgical Site Infections: A Meta-Analysis of Randomized Clinical Trials. Front Surg. 2022 Mar 25;9:855409. doi: 10.3389/fsurg.2022.855409. eCollection 2022. PMID 35402490
- [Background] Colunga-Lozano LE, Gonzalez Torres FJ, Delgado-Figueroa N, Gonzalez-Padilla DA, Hernandez AV, Roman Y, Cuello-Garcia CA. Sliding scale insulin for non-critically ill hospitalised adults with diabetes mellitus. Cochrane Database Syst Rev. 2018 Nov 29;11(11):CD011296. doi: 10.1002/14651858.CD011296.pub2. PMID 30488948
- [Background] Okabayashi T, Shima Y, Sumiyoshi T, Kozuki A, Tokumaru T, Iiyama T, Sugimoto T, Kobayashi M, Yokoyama M, Hanazaki K. Intensive versus intermediate glucose control in surgical intensive care unit patients. Diabetes Care. 2014 Jun;37(6):1516-24. doi: 10.2337/dc13-1771. Epub 2014 Mar 12. PMID 24623024
- [Background] Yuan J, Liu T, Zhang X, Si Y, Ye Y, Zhao C, Wang Q, Shen X. Intensive Versus Conventional Glycemic Control in Patients with Diabetes During Enteral Nutrition After Gastrectomy. J Gastrointest Surg. 2015 Aug;19(8):1553-8. doi: 10.1007/s11605-015-2871-7. Epub 2015 Jun 18. PMID 26084869
- [Background] Umpierrez GE, Smiley D, Zisman A, Prieto LM, Palacio A, Ceron M, Puig A, Mejia R. Randomized study of basal-bolus insulin therapy in the inpatient management of patients with type 2 diabetes (RABBIT 2 trial). Diabetes Care. 2007 Sep;30(9):2181-6. doi: 10.2337/dc07-0295. Epub 2007 May 18. PMID 17513708
- [Background] Migdal AL, Fortin-Leung C, Pasquel F, Wang H, Peng L, Umpierrez GE. Inpatient Glycemic Control With Sliding Scale Insulin in Noncritical Patients With Type 2 Diabetes: Who Can Slide? J Hosp Med. 2021 Aug;16(8):462-468. doi: 10.12788/jhm.3654. PMID 34328842
- [Background] Korytkowski MT, Muniyappa R, Antinori-Lent K, Donihi AC, Drincic AT, Hirsch IB, Luger A, McDonnell ME, Murad MH, Nielsen C, Pegg C, Rushakoff RJ, Santesso N, Umpierrez GE. Management of Hyperglycemia in Hospitalized Adult Patients in Non-Critical Care Settings: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2022 Jul 14;107(8):2101-2128. doi: 10.1210/clinem/dgac278. PMID 35690958